CLINICAL TRIAL: NCT01222806
Title: Pilot Study of Repetitive Transcranial Magnetic Stimulation (rTMS) in Cocaine Craving
Brief Title: Pilot Study of Repetitive Transcranial Magnetic Stimulation in Cocaine Craving
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 999911442; 11-DA-N442
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2013-05-02

CONDITIONS: Cocaine Use
Keywords: Functional Magnetic Resonance Imaging (fMRI); Cocaine; Cue-Induced Craving; Repetitive TMS (rTMS); Cocaine Craving
MeSH Terms: interventions — Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation

SUMMARY:
Background:

- Cocaine addiction is often difficult to treat, particularly because exposure to others using cocaine or to pictures of cocaine may evoke cocaine craving and lead a person to resume cocaine use after having quit. Breaking this link with cocaine craving might improve treatment for cocaine addiction. Research suggests that repetitive pulses of transcranial magnetic stimulation (rTMS) applied to the skull can change nerve cell firing in the brain. rTMS was recently approved as a treatment for depression, and is being studied as a way to reduce drug craving. However, because only a few small studies have looked at the effects of rTMS on cocaine craving, more research is needed on whether it is effective in reducing cocaine craving and use in individuals who currently use cocaine on a regular basis.

Objectives:

- To determine whether transcranial magnetic stimulation can lower craving for cocaine when given in connection with cocaine-related images.

Eligibility:

- Individuals at least 18 years of age who have used cocaine for at least 2 years and currently using at least 3 times per week.

Design:

* This study involves an initial screening visit, two brain imaging sessions, five rTMS sessions, and two follow-up visits.
* Participants will be screened with a medical history, physical examination, urine samples, questions about drug use history and previous efforts to quit, and tests for breath alcohol and nicotine levels.
* Participants will have two magnetic resonance imaging (MRI) scan sessions: one baseline scanning session before starting their rTMS sessions and a second scanning session after their last rTMS session . Part of each scanning session involves functional MRI (fMRI) scans. During the fMRI scans, participants will look at pictures related to cocaine use and pictures that are not related to cocaine use. Participants will also perform a simple decision task during the scans.
* Participants will have five rTMS sessions, one per day for 5 days in a row. Each session will last 1 to 2 hours. Participants will have either real or sham (simulated) rTMS while looking at pictures that may or may not be related to cocaine use, and will also perform a simple decision task that is the same as the one given during the MRI scans. The decision as to whether participants get real or sham rTMS will be made by chance. Neither the participants nor the investigators will know which type the participants are getting. - Participants will have two follow-up visits one and two weeks after their last rTMS session. At each visit they will be checked for cocaine and other substance use and for possible side-effects from rTMS.

DETAILED DESCRIPTION:
Primary objective: Repetitive transcranial magnetic stimulation (rTMS) provides a non-invasive means of altering brain neural activity. This pilot study will test whether 5 days of rTMS reduces cue-induced cocaine craving and cocaine use in cocaine users.

Hypothesis: We predict that active rTMS will significantly lower craving for cocaine compared with sham rTMS.

Study population: Thirty healthy adult cocaine users (for at least 2 years, currently averaging at least 3 times weekly) with no other major psychiatric disorders except nicotine dependence (DSM IV criteria) will be recruited from the community.

Design: Following a baseline phase to evaluate subject characteristics, subjects will be randomly assigned to receive 5 days of active or sham rTMS treatment. rTMS at 1 Hz and strength 120% of the motor threshold will be applied to the dorsolateral prefrontal cortex (DLPFC) using an H-coil (HADD version) contained in a helmet, beginning 1 second before presentation of a cocaine-associated visual cue and lasting for 30 seconds. Brain site localization will use a computerized navigation system based on structural MRI scans obtained before the first session. Each treatment session (lasting around 31 minutes) will consist of 54 trials (cue presentations): 36 with cocaine-associated cues and 9 each with non-drug-associated positive or neutral cues. No rTMS will be administered with the non-cocaine-associated cues. Subjects return for follow-up assessments one and two weeks after the final rTMS session.

Outcome measures: The primary outcome measure will be cocaine craving assessed by 100-mm visual analog scales before and after every TMS treatment and at one- and two week follow-up. Secondary outcome measures will be the 14-item Cocaine Craving Questionnaire, self-reported cocaine use, and urine drug testing at each rTMS session and follow-up visit, and changes in regional brain responses to cocaine-associated visual cues assessed by fMRI done before and after the 5 rTMS sessions.

Benefits: There is no direct benefit to individual subjects. The future benefit to society may be development of better methods for treatment of cocaine addiction.

Risks: The primary risks from rTMS are transient headache, scalp discomfort, decreased spatial recognition memory, and hearing loss (minimized by wearing ear plugs). Seizures are very rare when rTMS is administered within accepted safety guidelines and individuals at increased risk of seizures are excluded. The risk of inducing a manic episode is minimized by excluding individuals with a history of non-drug-induced mania/hypomania.

ELIGIBILITY:
-INCLUSION CRITERIA:

i) Eighteen to sixty-five years of age

ii) Cocaine user for at least 2 years, currently averaging at least 3 times weekly, with period of continuous abstinence no longer than one month within the past year

iii) Reading level of at least 6th grade, based on the Wide Range Achievement Test (WRAT)

iv) Ability to give valid informed consent

v) Right-handed

vi) If the subject is female and of childbearing potential, she agrees to use a medically acceptable form of contraception, and not become pregnant for the duration of the study. A woman is considered of childbearing potential unless post-menopausal or surgically sterilized. Female patients of childbearing potential must use either: (1) contraceptive pill or IUD or depot hormonal preparation (ring, injection, implant); and/or (2) a barrier method of contraception such as diaphragm, sponge with spermicide, or condom.

Contraceptive measures will be reviewed with female subjects at each visit prior to the rTMS treatment.

vii) Self-report experiencing cocaine craving when exposed to cocaine-associated cues

EXCLUSION CRITERIA:

i) Personal or first-degree family history of any clinically defined neurological disorder, including organic brain disease, epilepsy, stroke, brain lesions, or multiple sclerosis; or personal history of previous neurosurgery or head trauma that resulted in loss of consciousness.

ii) Cardiac pacemakers, neural stimulators, implantable defibrillator, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease, with intracranial implants (e.g. aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head that cannot be safely removed.

iii) Metal shrapnel or bullet in the head or body, including metal shavings.

iv) Current use of any investigational drug or of any medications with anti- or proconvulsive action, such as tricyclic antidepressants or neuroleptics (which lower seizure threshold).

v) Increased intracranial pressure (lowers seizure threshold)

vi) Lifetime history of major depressive disorder, schizophrenia, bipolar disorder, mania, or hypomania

vii) History of myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, or any heart condition currently under medical care.

viii) Pregnant or nursing women or women with reproductive potential not using an acceptable form of contraception.

ix) Any history of seizure

x) Current dependence (DSM-IV criteria) on substances other than cocaine and/or nicotine.

xi) Claustrophobia making them unable to tolerate lying in the MRI scanner.

xii) History of HIV infection or positive HIV antibody test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10-11; Study Completion 2013-05-02 (Actual)

PRIMARY OUTCOMES:
Cocaine Craving: cocaine craving questionnaire, visual-analogue scales | 2 weeks

SECONDARY OUTCOMES:
Cocaine Use: urine drug tests, self-report | 2 weeks
Side-Effects: side-effect checklist | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David A Gorelick, M.D., Principal Investigator — National Institute on Drug Abuse (NIDA)

REFERENCES:
- [Background] Agosti V, Nunes E, Ocepeck-Welikson K. Patient factors related to early attrition from an outpatient cocaine research clinic. Am J Drug Alcohol Abuse. 1996 Feb;22(1):29-39. doi: 10.3109/00952999609001643. PMID 8651143
- [Background] Allen EA, Pasley BN, Duong T, Freeman RD. Transcranial magnetic stimulation elicits coupled neural and hemodynamic consequences. Science. 2007 Sep 28;317(5846):1918-21. doi: 10.1126/science.1146426. PMID 17901333
- [Background] Bestmann S, Baudewig J, Siebner HR, Rothwell JC, Frahm J. Functional MRI of the immediate impact of transcranial magnetic stimulation on cortical and subcortical motor circuits. Eur J Neurosci. 2004 Apr;19(7):1950-62. doi: 10.1111/j.1460-9568.2004.03277.x. PMID 15078569